CLINICAL TRIAL: NCT00745641
Title: Effect of Abdominal X-ray Computed Tomography Examination on the Blood Reactive Oxygen Species Level
Brief Title: Abdominal Computed Tomography and the Blood Reactive Oxygen Species Level
Status: Withdrawn | Type: Observational
Why Stopped: because of the presence of unexpected administrative barrier to interfere the collection of case
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Zei-Shung Huang, associate professor, Department of Internal Medicine, NTUH, National Taiwan University Hospital
Other Study IDs: 200807056R
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-03

CONDITIONS: Radiation Injury
Keywords: radiation injury; computed tomography; reactive oxygen species; free radicals
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — only peripheral blood will be collected for measurement of reactive oxygen species.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Sixty patients with abdominal illness and scheduled abdominal X-ray computed tomography examination will be included.

SUMMARY:
The clinically widely used X-ray computed tomography examination has a low-grade radiation effect and recently has attracted much attention concerning the possible adverse effects of radiation on human body [ref. 1-5]. The radiation is harmful to human tissues and cells mainly because it can interact with water (which makes up to 80% of cells) to generate reactive oxygen species (ROS), especially the formation of hydroxyl radicals. So far as we can reach, there is no report concerning the relation between X-ray computed tomography examination and the blood ROS level. Therefore, we wish to conduct this study to clarify if the routinely applied abdominal X-ray computed tomography examination may induce a higher level of ROS in the peripheral blood.

Study subjects will be patients who are admitted to our hospital because of abdominal diseases that need to receive abdominal X-ray computed tomography examination for diagnosis. In total, sixty cases will be enrolled for the study. The formal consent will be delivered and explained to the patients and families several hours before the performance of abdominal X-ray computed tomography. The formal consent will be retrieved and then the peripheral blood will be sampled just before the performance of computed tomography.ROS level in the sampled peripheral blood, before and after the performance of abdominal X-ray computed tomography, will be measured, compared, and analyzed. Totally 120 blood samples, including 60 samples just before and 60 samples 2 hours after the performance of computed tomography, will be collected from 60 study subjects within 5 months (August 10 ~ December 30, 2008). Reactive oxygen species（ROS）levels will be measured by a chemiluminescence (CL) analysing system (CLD-110, Tohoku Electronic Industrial, Sendai, Japan).

ELIGIBILITY:
Inclusion Criteria:

* patients with abdominal illness that needs a computed tomography examination

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with abdominal illness that needs a computed tomography examination
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zei-Shung Huang, MD, PhD, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan